CLINICAL TRIAL: NCT05059314
Title: Effects Of Moderate Physical Activity On Hb, Physical Fitness And Psychological Well Being In Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/00929 Rabbya Kausar
Record Dates: First submitted 2021-03-12; First posted 2021-09-28 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Anemia; Quality of Life
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant
Masking Description: According to study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): 1. Warm up and cool down
  2. Brisk walk (30 mintues each session per week 5 days)
  3. Week 1 to 6
  Interventions: Other: Brisk walking (moderate physical activity)
- Control group (No Intervention): Routine activity

INTERVENTIONS:
Other: Brisk walking (moderate physical activity) — 1. Warm up and cool down
  2. Brisk walk (30 mintues each session per week 5 days)
  3. Week 1 to 6
  Other Names: Moderate physical activity
  Arms: Interventional group

SUMMARY:
The study is design To determine the effectiveness of moderate physical activity on Hb, Physical fitness and psychological well-being in females.

DETAILED DESCRIPTION:
The majority of literature showed that level of physical activity is associated with Hb level. But there is paucity in the literature regarding the cause and effect relationship of PA and Hb. Literature shows lacking that there is any defined physical activity, which can affect the Hb concentration. According to literature, different studies conduct at Hb level in individuals with different diseases i.e. rheumatic arthritis, Diabetes mellitus etc. The aim of my study is to determining the cause and effect relationship of moderate physical activity on Hb level in healthy female population, one of the easiest moderate physical activity is brisk walk. Brisk walk is an aerobic exercise. People do get best physiological results of aerobic exercise with intensity of exercise 60-70% of the maximum pulse with longer time duration as well as increase frequency of exercise, which increase no of hemoglobin level due to this need more oxygen to performing physical activity in return basal metabolic rate increases and achieve physical fitness and gain relieve from the psychological problems.

ELIGIBILITY:
Inclusion Criteria:

1. Female 2.18-25 years 3. Hb<12

Exclusion Criteria:

1. Lower limb musculoskeletal injury
2. Any head Injury or trauma in past 6 months.
3. Any neurological or musculoskeletal condition
4. Acute or chronic infections diseases

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self representation of gender identity
Enrollment: 22 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Hemoglobin level concentration | 6 week
  Hemoglobin is a protein in red blood cells that carries iron. In adults,In study hemoglobin level will be measured in healthy females which will be less than 12.
Physical activity readiness questionnaire (PAR-Q) | 6 week
  The Physical Activity Readiness Questionnaire (PAR-Q) is a common method of uncovering health and lifestyle issues prior to an exercise programme starting. The questionnaire is short and easy to administer and reveals any family history of illness.
Physical Fitness Test ( 12-minute run test) | 6 week
  The 12-minute run fitness test as an easy way to measure aerobic fitness .The Cooper 12-minute run test requires the person being tested to run or walk as far as possible in a 12-minute period. The objective of the test is to measure the maximum distance covered by the individual during the 12-minute period
Physical Fitness Test( Shuttle run test) | 6 weeks
  Shuttle Run is a test of agility, in which the participant runs back and forth between two parallel lines as fast as possible.
Physical Fitness Test(Sit and reach test) | 6 weeks
  The sit and reach test is a common measure of flexibility, and specifically measures the flexibility of the lower back and hamstring muscles.
Physical fitness test(lateral plyometric test) | 6 weeks
  Lateral plyometric jumps are advanced exercises that can be used to develop power and agility
Physical fitness test(Push-ups) | 6 weeks
  The upper body muscles that come into play in the pushup are the deltoids of the shoulders, the pectoral muscles of the chest, the triceps and biceps of the upper arm, and the erector spinae of the back.
Perceived stress scale (PSS) | 6 weeks
  The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful.
International physical activity Questionaire (IPAQ) | 6 weeks
  We are interested in finding out about the kinds of physical activities that people do as part of their everyday lives. The questions will ask you about the time you spent being physically active in the last 7 days.
Quality of life SF-12 scale | 6 weeks
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
VO2max | 6 weeks
  V̇O₂ max is the maximum rate of oxygen consumption measured during incremental exercise; that is, exercise of increasing intensity. The name is derived from three abbreviations: "V̇" for volume, "O₂" for oxygen, and "max" for maximum.

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmad Awan, PhD, Principal Investigator — Riphah International University
Locations (1):
- Pakistan, Islamabad, Pakistan/Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No